CLINICAL TRIAL: NCT01903733
Title: AN OPEN-LABEL BOSUTINIB TREATMENT EXTENSION STUDY FOR SUBJECTS WITH CHRONIC MYELOID LEUKEMIA (CML) WHO HAVE PREVIOUSLY PARTICIPATED IN BOSUTINIB STUDIES B1871006 OR B1871008
Brief Title: Bosutinib Treatment Extension Study Only For Subjects With Chronic Myeloid Leukemia (CML) Who Have Previously Participated In Bosutinib Studies B1871006 Or B1871008
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: B1871040; 2013-000691-15 (EudraCT Number)
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-06

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Subjects; Chronic Myeloid Leukemia; CML; Bosutinib; Extension
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bosutinib — The starting bosutinib dose is 500 mg once daily, however the dose can vary from 300 mg to 600 mg.

SUMMARY:
The objective of the study is to provide long term access to bosutinib treatment and assess long term safety, tolerability and duration of clinical benefit, without any formal hypothesis testing; therefore, there is no formal primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects previously participating in two specific studies are eligible to enroll into this study. Enrollment is not open to subjects if not previously enrolled in studies B1871006 or B1871008.

Exclusion Criteria:

* All subjects are excluded unless previously participating in studies B1871006 or B1871008.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2013-08-28 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (90):
- United States (13):
  - Orlando Health, Inc, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northside Hospital Inc., - GCS/Northside, Atlanta, Georgia
  - Northside Hospital, Inc. - Central Research Department, Atlanta, Georgia
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Rcca Md,Llc, Bethesda, Maryland
  - Hudson Valley Hematology and Oncology Associates, Hawthorne, New York
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas
- Argentina (3):
  - Instituto Medico Especializado Alexander Fleming, Cd. Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de la Plata, La Plata, Buenos Aires
  - Hospital Dr. Jose Ramon Vidal, Corrientes
- Australia (2):
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- GHDC (Grand Hopital de Charleroi), Charleroi, Belgium
- Brazil (2):
  - Universidade Estadual de Campinas / Centro de Hematologia e Hemoterapia, Campinas, São Paulo
  - Faculdade de Medicina do ABC - Centro de Estudos e Pesquisa em Hematologia e Oncologia (CEPHO), Santo André, São Paulo
- Canada (4):
  - Alberta Health Services - Department of Medical Oncology - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sir Mortimer B. Davis-Jewish General Hospital, Montreal, Quebec
- Chile (2):
  - Instituto Oncologico, Clinica Renaca, Reñaca, Región de Valparaíso
  - Instituto Oncologico, Reñaca, Región de Valparaíso
- China (5):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Chinese People's Liberation Army General Hospital, Beijing
  - Ruijin Hospital- Shanghai Jiaotong University School of Medicine, Shanghai
  - Blood Disease Hospital, Chinese Academy of Medical Science & Peking Union Medical College, Tianjin
- Fundacion Santa Fe de Bogota, Bogota, Cundinamarca, Colombia
- Helsingin Yliopistollinen Keskussairaala, Hematologian poliklinikka, Helsinki, Finland
- France (5):
  - CHU de CAEN, Caen
  - CHU Hotel Dieu - Service Hematologie, Nantes
  - CHU de Poitiers, Poitiers
  - CHU Poitiers, Poitiers
  - Strasbourg Oncologie Liberale -Centre de Radiotherapie, Clinique Ste Anne, Strasbourg
- Hong Kong (2):
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan
  - Department of Medicine & Therapeutics, Prince of Wales Hospital, Shatin, New Territories
- Hungary (2):
  - Egyesitett Szent Istvan es Szent Laszlo Korhaz-Rendelointezet, Budapest
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Belgyogyaszati Osztaly, Kaposvár
- Christian Medical College. Vellore, Vellore, Tamil Nadu, India
- Italy (4):
  - A.O.U. Policlinico S.Orsola Malpighi, Bologna, BO
  - ASST Monza - Ospedale san Gerardo, Monza, Monza and Brianza
  - A.O.U. San Luigi Gonzaga di Orbassano, Orbassano, TO
  - Ospedale S. Eugenio - UOC Ematologia, Roma
- Japan (8):
  - Toyohashi Municipal Hospital, Toyohashi, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Hamamatsu University School of Medicine University Hospital, Hamamatsu, Shizuoka
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Tokyo
- Riga East Clinical University Hospital, Riga, Latvia
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - University Medical Center Groningen, Department of Hematology, Groningen
- Unidad de Investigacion de Hematologia - Hospital Nacional Edgardo Rebagliati Martins, Lima, Peru
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Samodzielny Publiczny Szpital Kliniczny nr 1 w Lublinie, Lublin
- Russia (8):
  - State Budgetary Institution of Healthcare of Sverdlovsk Region, Yekaterinburg, Sverdlovsk Oblast
  - Federal State-Funded Institution National Research Center of Hematology of the Ministry of, Moscow
  - State Budgetary Institution of Rostov Region - Rostov Regional Clinical Hospital, Rostov-on-Don
  - State Budgetary Educational Institution of Higher Professional Education, Rostov-on-Don
  - State Budgetary Institution of Healthcare - Leningrad Regional Clinical Hospital, Saint Petersburg
  - Clinic "Institute of Pediatric Oncology, Hematology and Transplantation n.a. R.M. Gorbachova", Saint Petersburg
  - Federal State Budgetary Institution "Federal Almazov Medical Research Centre", Saint Petersburg
  - State Budgetary Institution of Healthcare Samara Regional Clinical Hospital n.a. V.D. Seredavin, Samara
- Singapore General Hospital, Singapore, Singapore
- Wits Clinical Research-Chris Hani Baragwanath Hospital, Soweto, Gauteng, South Africa
- The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, South Korea
- Spain (6):
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Madrid Sanchinarro, Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clinico Universitario De Valencia (CHUV), Valencia
- Division of Hematology, Department of Medicine, Faculty of Medicine, Siriraj Hospital,, Bangkok, Thailand
- Turkey (Türkiye) (2):
  - Gaziantep Universitesi Tip Fakultesi Sahinbey Uygulama ve Arastirma Hastanesi, Gaziantep, Sehit Kamil
  - Hacettepe Universitesi Tip Fakultesi, Ankara
- Ukraine (5):
  - Municipal Institution "Cherkasy Regional Oncology Dispensary", Cherkasy
  - MI "Dnipropetrovsk City Multi-field Clinical Hospital #4" of DRC Hematology Center, Dnipropetrovsk
  - State Institution "National Research Center for Radiation Medicine of the National Academy of, Kyiv
  - Kyiv City Clinical Hospital #9, SI "Institute of Hematology and Transfusiology of NAMS of Ukraine", Kyiv
  - State Institution "Institute of Blood Pathology and Transfusion Medicine of, Lviv
- United Kingdom (2):
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottinhgam

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Takahashi N, Cortes JE, Sakaida E, Ishizawa K, Ono T, Doki N, Matsumura I, Garcia-Gutierrez V, Rosti G, Ono C, Ohkura M, Tanetsugu Y, Viqueira A, Brummendorf TH. Safety profile of bosutinib in Japanese versus non-Japanese patients with chronic myeloid leukemia: a pooled analysis. Int J Hematol. 2022 Jun;115(6):838-851. doi: 10.1007/s12185-022-03314-y. Epub 2022 Mar 2. PMID 35235189
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1871040&StudyName=An%20Open-label%20Bosutinib%20Treatment%20Extension%20Study%20For%20Subjects%20With%20Chronic%20Myeloid%20Leukemia%20%28cml%29%20Who%20Have%20Previously%20Participated%20In%20Bosutinib%20Studies%20B1871006%20Or%20B1871008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was offered to participants randomized to bosutinib arm in B1871008 (NCT00574873) or dosed with bosutinib in B1871006 (NCT00261846). Participants enrolled in this study were who in any of the parent studies (B1871008 or B1871006) at time of protocol approval 1) receiving bosutinib, benefiting per investigator, 2) discontinued bosutinib, being followed-up,3) completed parent study. Per enrolment criteria, 281 participants were enrolled in this study and 21 participants were from China.
Pre-assignment Details: Per protocol data from 2 parent studies were combined with data from this study (B1871040) for all analyses. Reporting arms were based on parent study, disease phase and line of therapy (CP1L,CP2L,CP3L/CP4L,ADV).The B1871040 data from 21 participants enrolled in China were not included in results because the Human Genetics Resources Administration of China did not approve the use of the data in accordance with its regulations. This data has been excluded from all our analyses.
Groups:
- Bosutinib, CP1L: Participants from B1871008 with Philadelphia chromosome-positive (Ph+) chronic phase 1st line (CP1L) chronic myeloid leukemia (CML) who either continued to receive the same bosutinib dose as at the time of completion of B1871008 or continued to be followed for survival. Dose for bosutinib was 500 milligram (mg) orally once daily (adjusted dose varied from 200 mg to 600 mg once daily). Treatment continued until the end of the study, disease progression, unacceptable toxicity, death, withdrawal of consent or study discontinuation whichever occurred first. Follow-up continued till end of the study or death due to any cause whichever occurred first. Participants remained in this study, either for treatment or for follow-up, until the last participant enrolled in 1 of the parent studies reached 10 years of follow-up, as calculated from the date of his/her first dose of bosutinib administered in parent study.
- Bosutinib, CP2L: Participants from B1871006 with Ph+ chronic phase 2nd line (CP2L) CML who were resistant or intolerant to imatinib either continued to receive the same bosutinib dose as at the time of completion of B1871006 or continued to be followed for survival. Dose for bosutinib was 500 mg orally once daily (adjusted dose varied from 200 mg to 600 mg once daily). Treatment continued until the end of the study, disease progression, unacceptable toxicity, death, withdrawal of consent or study discontinuation whichever occurred first. Follow-up continued till end of the study or death due to any cause whichever occurred first. Participants remained in this study, either for treatment or for follow-up, until the last participant enrolled in 1 of the parent studies reached 10 years of follow-up, as calculated from the date of his/her first dose of bosutinib administered in parent study.
- Bosutinib, CP3L/CP4L: Participants from B1871006 with Ph+ chronic phase 3rd line (CP3L)/4th line (CP4L) CML who were resistant or intolerant to imatinib and resistant or intolerant to dasatinib and/or nilotinib either continued to receive the same bosutinib dose as at the time of completion of B1871006 or continued to be followed for survival. Dose for bosutinib was 500 mg orally once daily (adjusted dose varied from 200 mg to 600 mg once daily). Treatment continued until the end of the study, disease progression, unacceptable toxicity, death, withdrawal of consent or study discontinuation whichever occurred first. Follow-up continued till end of the study or death due to any cause whichever occurred first. Participants remained in this study, either for treatment or for follow-up, until the last participant enrolled in 1 of the parent studies reached 10 years of follow-up, as calculated from the date of his/her first dose of bosutinib administered in parent study.
- Bosutinib, ADV: Advanced (ADV) participants from B1871006 with Ph+ accelerated phase (AP), blast phase (BP) CML, Ph+ acute lymphoblastic leukemia (ALL) and resistant or intolerant to imatinib only or resistant or intolerant to imatinib and at least 1 additional tyrosine kinase inhibitor (TKI) including dasatinib and/or nilotinib who either continued to receive the same bosutinib dose as at the time of completion of B1871008 or continued to be followed for survival. Dose for bosutinib was 500 mg orally once daily (adjusted dose varied from 200 mg to 600 mg once daily). Treatment continued until the end of the study, disease progression, unacceptable toxicity, death, withdrawal of consent or study discontinuation whichever occurred first. Follow-up continued till end of the study or death due to any cause whichever occurred first. Participants remained in this study, either for treatment or for follow-up, until the last participant enrolled in 1 of the parent studies reached 10 years of follow-up, as calculated from the date of his/her first dose of bosutinib administered in parent study.
Period: Overall Study
Arm/Group | Bosutinib, CP1L | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV
Started | 250 | 284 | 119 | 167
Full Analysis Set ((participants randomized to bosutinib arm in B1871008 and all dosed participants in B1871006)) | 250 | 284 | 119 | 167
Safety Analysis Set ((all dosed participants in B1871008 and B1871006)) | 248 | 284 | 119 | 167
Enrolled in B1871040 | 124 | 90 | 28 | 18
Treated in B1871040 | 98 | 69 | 13 | 8
Completed | 144 | 158 | 58 | 48
Not Completed | 106 | 126 | 61 | 119
Not completed — Death | 23 | 54 | 30 | 98
Not completed — Participant refused further follow-up | 35 | 38 | 13 | 9
Not completed — Lost to Follow-up | 18 | 19 | 6 | 9
Not completed — Other | 10 | 15 | 12 | 3
Not completed — Missing | 2 | 0 | 0 | 0
Not completed — Investigator request | 18 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants randomized to the bosutinib arm from B1871008 and all dosed participants from B1871006.
Groups:
- Bosutinib, CP1L: Participants from B1871008 with Philadelphia chromosome-positive (Ph+) chronic phase 1st line (CP1L) chronic myeloid leukemia (CML).
- Bosutinib, CP2L: Participants from B1871006 with Ph+ chronic phase 2nd line (CP2L) CML who were resistant or intolerant to imatinib.
- Bosutinib, CP3L/CP4L: Participants from B1871006 with Ph+ chronic phase 3rd line (CP3L)/4th line (CP4L) CML who were resistant or intolerant to imatinib and resistant or intolerant to dasatinib and/or nilotinib.
- Bosutinib, ADV: Participants from B1871006 with Ph+ accelerated phase (AP), blast phase (BP) CML or Ph+ acute lymphoblastic leukemia (ALL) and resistant or intolerant to imatinib only or resistant and intolerant to imatinib and at least 1 additional tyrosine kinase inhibitor (TKI) including dasatinib and/or nilotinib.
- Total: Total of all reporting groups
Arm/Group | Bosutinib, CP1L | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV | Total
Number analyzed (Participants) | 250 | 284 | 119 | 167 | 820
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.9 (14.4) | 51.9 (15.1) | 55.1 (13.0) | 50.1 (15.4) | 50.8 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 135 | 66 | 69 | 371
  Male | 149 | 149 | 53 | 98 | 449
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 83 | 61 | 15 | 37 | 196
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 16 | 6 | 19 | 43
  White | 160 | 186 | 87 | 102 | 535
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 20 | 11 | 9 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) Based on National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) (Version 3.0)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening (immediate risk of death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions), resulted in congenital anomaly/birth defect. Treatment-emergent adverse events were defined as any event increasing in severity from baseline or any new event started during bosutinib therapy or within 30 days of the last dose of study drug.
Time Frame: From first dose of drug up to 30 days after last dose (up to approximately 14 years)
Population: Safety analysis set included all dosed participants for both B1871006 and B1871008.
Measure: Count of Participants; unit: Participants
Groups:
- Bosutinib, Total: Participants from B1871008 CP1L cohort and B1871006 CP2L, CP3L/CP4L and ADV cohorts.
Arm/Group | Bosutinib, CP1L | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV | Bosutinib, Total
Number analyzed (Participants) | 248 | 284 | 119 | 167 | 818
Participants
  Treatment-Emergent AEs | 241 | 283 | 119 | 165 | 808
  Treatment-emergent SAEs | 102 | 124 | 44 | 98 | 368

2. Primary Outcome: Number of Participants With Grade 3 or 4 Treatment-Emergent Adverse Events (AEs) Based on National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) (Version 3.0)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs were assessed according to severity grading based on NCI CTCAE version 3.0. Grade 1 =mild; Grade 2 =moderate; Grade 3 =severe or medically significant but not immediately life-threatening, hospitalization or prolongation of hospitalization indicated; Grade 4 =life-threatening or disabling, urgent intervention indicated; Grade 5 =death. Treatment-emergent adverse events were defined as any event increasing in severity from baseline or any new event started during bosutinib therapy or within 30 days of the last dose of study drug.
Time Frame: From first dose of drug up to 30 days after last dose (up to approximately 14 years)
Population: Safety analysis set included all dosed participants for both B1871006 and B1871008.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib, CP1L | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV | Bosutinib, Total
Number analyzed (Participants) | 248 | 284 | 119 | 167 | 818
Participants | 191 | 223 | 84 | 144 | 642

3. Primary Outcome: Number of Participants With Treatment-Emergent Treatment Related Adverse Events (AEs) Based on National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) (Version 3.0)
Description: An AE was any untoward medical occurrence in a participant who received study drug. Treatment-emergent adverse events were defined as any event increasing in severity from baseline or any new event started during bosutinib therapy or within 30 days of the last dose of study drug. Related TEAEs were those AEs who were related to the study treatment as judged by the investigator.
Time Frame: From first dose of drug up to 30 days after last dose (up to approximately 14 years)
Population: Safety analysis set included all dosed participants for both B1871006 and B1871008.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib, CP1L | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV | Bosutinib, Total
Number analyzed (Participants) | 248 | 284 | 119 | 167 | 818
Participants | 235 | 282 | 119 | 161 | 797

4. Primary Outcome: Number of Participants With Laboratory Test Abnormalities Based on National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) (Version 4.03)
Description: Laboratory parameters included Chemistry: high alkaline phosphatase; high alanine aminotransferase; high aspartate aminotransferase; high blood bilirubin; high creatinine. Hematology: absolute neutrophils count decreased; anemia; platelet count decreased; white blood cells (WBC) decreased. Abnormalities in laboratory tests were graded per NCI CTCAE version 4.03 as Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling.
Time Frame: From first dose of drug up to 30 days after last dose (up to approximately 14 years)
Population: Safety analysis set included all dosed participants for both B1871006 and B1871008.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib, CP1L | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV | Bosutinib, Total
Number analyzed (Participants) | 248 | 284 | 119 | 167 | 818
Participants
  Grade 1 | 45 | 59 | 28 | 18 | 150
  Grade 2 | 86 | 80 | 39 | 24 | 229
  Grade 3 | 84 | 102 | 27 | 41 | 254
  Grade 4 | 33 | 42 | 23 | 82 | 180

5. Primary Outcome: Number of Participants With Adverse Events as Reason for Treatment Discontinuation
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: From first dose of drug up to 30 days after last dose (up to approximately 14 years)
Population: Safety analysis set included all dosed participants for both B1871006 and B1871008.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib, CP1L | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV | Bosutinib, Total
Number analyzed (Participants) | 248 | 284 | 119 | 167 | 818
Participants | 84 | 79 | 37 | 32 | 232

6. Primary Outcome: Number of Participants With Diarrhea After Switch From Bosutinib Clinical Formulation to Bosutinib Commercial Formulation
Description: The incidence of diarrhea was collected and analyzed before and after the switch from the clinical formulation of bosutinib to the commercial formulation of bosutinib.
Time Frame: Last 6 months on clinical formulation and first 6 months on commercial formulation
Population: Safety analysis set included all dosed participants for both B1871006 and B1871008. Here, 'Overall number of participants analyzed'= participants evaluable for this outcome measure who received commercial formulation.
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib, CP1L | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV | Bosutinib, Total
Number analyzed (Participants) | 119 | 82 | 13 | 8 | 222
Participants
  Clinical formulation (last 6 months) | 25 | 22 | 3 | 5 | 55
  Commercial formulation (first 6 months) | 34 | 27 | 4 | 5 | 70

7. Primary Outcome: Number of Participants With Breakpoint Cluster Region Abelson Protooncogene (BCR-ABL) Mutations Present at Time of Bosutinib Treatment Discontinuation
Description: BCR-ABL is a gene resulting from the 9:22 chromosomal translocation (Philadelphia chromosome). In this outcome measure, the number of participants who had emergent mutation or new BCR-ABL mutations (participants who had a post-baseline mutation which was not present at baseline) were reported.
Time Frame: Post-baseline on Day 1 (maximum up to 14 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Bosutinib, CP1L | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV
Number analyzed (Participants) | 250 | 284 | 119 | 167
Participants | 7 | 28 | 13 | 14

8. Primary Outcome: Overall Survival (OS) Rate at Year 10
Description: OS was defined as the time from randomization (B1871008) and time from first dose (B1871006) to the occurrence of death due to any cause or censoring. Kaplan-Meier analysis was used for determination of OS. Percentage of participants who were alive were estimated in this outcome measure.
Time Frame: Year 10
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib, CP1L | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV
Number analyzed (Participants) | 250 | 284 | 119 | 167
percentage of participants | 88.2 [83.3 to 93.2] | 71.5 [64.4 to 78.7] | 60.4 [47.2 to 73.7] | 34.2 [25.0 to 43.4]

9. Primary Outcome: Plasma Steady-State Trough Concentrations (Ctrough) of Bosutinib
Description: Ctrough refers to plasma concentration of bosutinib observed just before treatment administration.
Time Frame: One pre-dose sample was collected at the first scheduled visit (after approval and implementation of protocol amendment 1) following at least 2 weeks of uninterrupted dosing at the same dose level
Population: The pharmacokinetic (PK) analysis set included participants who received at least 1 dose of bosutinib and had 1 reported bosutinib concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Groups:
- Bosutinib 200 mg: Participants received uninterrupted once daily oral 200 mg dose of bosutinib for at least 2 weeks in study B1871040.
- Bosutinib 300 mg: Participants received uninterrupted once daily oral 300 mg dose of bosutinib for at least 2 weeks in study B1871040.
- Bosutinib 400 mg: Participants received uninterrupted once daily oral 400 mg dose of bosutinib for at least 2 weeks in study B1871040.
- Bosutinib 500 mg: Participants received uninterrupted once daily oral 500 mg dose of bosutinib for at least 2 weeks in study B1871040.
- Bosutinib 600 mg: Participants received uninterrupted once daily oral 600 mg dose of bosutinib for at least 2 weeks in study B1871040.
Arm/Group | Bosutinib 200 mg | Bosutinib 300 mg | Bosutinib 400 mg | Bosutinib 500 mg | Bosutinib 600 mg
Number analyzed (Participants) | 6 | 28 | 23 | 69 | 8
nanogram per milliliter | 62.2 (31.3) | 62.0 (65.9) | 82.2 (53.2) | 93.3 (45.2) | 99.4 (78.2)

10. Primary Outcome: Kaplan-Meier Estimate of Probability of Maintaining Major Cytogenetic Response (MCyR) at Year 10: B1871006 Participants
Description: Cytogenetic response (CyR) is based on prevalence of Ph+ cells. Duration for MCyR: time from first response to confirmed loss, progression of disease, or on-treatment death due to any cause, or censoring analyzed for responders only. Confirmed loss was defined as 2 consecutive non-responses at least 28 days apart. MCyR was categorized as either complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR). Response was achieved when there was 0% (CCyR) or 1-35% (PCyR) Ph+ cells analyzed from conventional cytogenetics based on the analysis of 20 to 100 metaphases or <1% (CCyR) or 1-35% (PCyR) Ph+ cells analyzed from fluorescence in-situ hybridization (FISH) based on analysis of at least 200 nuclei. CCyR may be imputed on a specific date if an MMR or better is achieved and denoted on the CRF on that date for B1871040 study visits. The Kaplan-Meier analysis was used to analyze percentage of participants maintaining MCyR at Year 10.
Time Frame: Year 10
Population: The evaluable analysis set for cytogenetic population were those dosed participants from B1871006 with valid baseline efficacy assessment from B1871006 with >=20 metaphases or at least 1 Ph+ metaphase from baseline bone marrow cytogenetic assessment and who achieved MCyR (responders). "N"=evaluable participants. Data for this outcome measure was planned to be collected and analyzed for participants from B1871006 only and not for reporting arm "Bosutinib CP1L" (participants from B1871008).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV
Number analyzed (Participants) | 157 | 47 | 54
percentage of participants | 65.3 [56.6 to 74.0] | 55.3 [36.3 to 74.4] | 30.6 [16.4 to 44.7]

11. Primary Outcome: Kaplan-Meier Estimate of Probability of Maintaining Complete Cytogenetic Response (CCyR) at Year 10: B1871006 Participants
Description: Duration for CCyR was defined as time from first response to confirmed loss, progression of disease, or on-treatment death due to any cause, or censoring analyzed for responders only. Confirmed loss was defined as 2 consecutive assessments with >0 Ph+ metaphases or >=1% positive cells from FISH at least 28 days apart or progression or death. CCyR was achieved when there was 0% Ph+ cells analysed from conventional cytogenetics with 20 to 100 metaphases or <1% Ph+ cells analysed from FISH with at least 200 nuclei. CCyR may be imputed on a specific date if MMR or better is achieved and denoted on the CRF on that date for B1871040 study visits. The Kaplan-Meier analysis was used to analyze percentage of participants maintaining CCyR at Year 10.
Time Frame: Year 10
Population: The evaluable analysis set for cytogenetic population were those dosed participants from B1871006 with a valid baseline efficacy assessment from B1871006 with >=20 metaphases or at least 1 Ph+ metaphase from the baseline bone marrow cytogenetic assessment and who achieved CCyR (responders). "N"=evaluable participants. Data for this outcome measure was planned to be collected and analyzed for participants from B1871006 only and not for reporting arm "Bosutinib CP1L" (participants from B1871008).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV
Number analyzed (Participants) | 130 | 36 | 42
percentage of participants | 63.4 [54.0 to 72.8] | 40.8 [22.0 to 59.6] | 29.6 [14.6 to 44.7]

12. Primary Outcome: Kaplan-Meier Estimate of Probability of Maintaining Complete Hematologic Response (CHR) at Year 10: B1871006 Participants
Description: Duration for CHR was defined as time from first response to confirmed loss, progression of disease, or on-treatment death due to any cause, or censoring analyzed for responders only. Confirmed loss was defined as 2 consecutive non-responses at least 14 days apart. Complete hematologic response was considered when participants met all of the following criteria: White blood cells equal to or less than (<=) institutional upper limit of normal (ULN), no blasts or promyelocytes in blood, <20% basophils in blood, no extramedullary involvement (including hepatomegaly or splenomegaly), myelocytes and metamyelocytes <5% in blood, platelets <450*10^9 per liter (/L). The following were applicable only to advanced phase: <=5% bone marrow blasts, absolute neutrophil count >=1.0*10^9/L, platelets >=100*10^9/L. The Kaplan-Meier analysis was used to analyze percentage of participants maintaining CHR at Year 10.
Time Frame: Year 10
Population: The evaluable analysis set for hematologic population were those dosed participants from B1871006 with a valid baseline efficacy assessment from B1871006 and a valid baseline hematologic assessment and who achieved CHR (responders). "N"=evaluable participants. Data for this outcome measure was planned to be collected and analyzed for participants from B1871006 only and not for reporting arm "Bosutinib CP1L" (participants from B1871008).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV
Number analyzed (Participants) | 245 | 86 | 36
percentage of participants | 44.1 [35.2 to 52.9] | 45.1 [29.3 to 60.9] | NA [NA to NA] — The percentage and 95% CI was not estimable since BM blasts were not always assessed in later years for ADV participants.

13. Primary Outcome: Cumulative Incidence of Progression/Death Events at Year 10: B1871006 Participants
Description: Progression free survival (PFS):interval from date of first dose of bosutinib in parent study until earlier date of progression or death from any cause. Participants without events censored at last evaluation date. PD:evolution from CP (or return to CP for ADV participants) to AP or BP (on 2 consecutive assessments at least 1 week apart), evolution from AP to BP (on 2 consecutive assessments at least 1 week apart) and one of following conditions occurred after dose escalation or presence of AEs prohibiting dose escalation: for 2nd or later line, loss of MCyR (need at least 30% increase); for all lines of treatment, loss of CHR confirmed by 2 assessments >=2 weeks apart; for all lines of treatment, increasing WBC defined as doubling of WBC over a period of >=1 month with second WBC >20*10^9/L confirmed at least 1 week later. Percentage of participants with PFS/death events based on cumulative incidence method adjusting for competing event of treatment discontinuation without event.
Time Frame: Year 10
Population: The full analysis set from B1871006 included all dosed participants from the study B1871006. Data for this outcome measure was planned to be collected and analyzed for participants from B1871006 only and not for reporting arm "Bosutinib CP1L" (participants from B1871008).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV
Number analyzed (Participants) | 284 | 119 | 167
percentage of participants | 23.9 [19.5 to 29.5] | 26.9 [20.0 to 36.2] | 55.7 [48.6 to 63.8]

14. Primary Outcome: Cumulative Incidence of Rate of Transformation to Accelerated Phase (AP) or Blast Phase (BP) at Year 10: B1871006 Participants
Description: Time to transformation was defined as the time from first dose in the parent study to the first date of confirmed transformation to AP or BP. Confirmed transformation was defined as 2 consecutive assessments at least 1 week apart or 1 assessment confirmed by progression of disease or death. For participants without transformation, censorship was at the last evaluation date. Percentage of participants with time to transformation to AP/BP was reported based on cumulative incidence method adjusting for the competing risk of treatment discontinuation without the event.
Time Frame: Year 10
Population: The full analysis set from B1871006 included all dosed participants from the study B1871006. Data for this outcome measure was planned to be collected and analyzed for participants from B1871006 only and not for reporting arm "Bosutinib, CP1L" (participants from B1871008). For "Bosutinib ADV" reporting arm, data was analyzed for participants with AP who had BP transformation only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV
Number analyzed (Participants) | 284 | 119 | 79
percentage of participants | 5.3 [3.2 to 8.6] | 4.2 [1.8 to 9.9] | 3.8 [1.3 to 11.5]

ADVERSE EVENTS:
Time Frame: From first dose of study drug and up to 30 days after last dose (up to approximately 14 years)
Description: All-cause mortality: The total number of deaths during study, from randomization (B1871008)/first dose (B1871006) and up to the end of the study are reported for all treated participants and includes deaths which occurred after 30 days post last study drug dose. SAEs and other AEs: Analysis performed on safety set. Data from the 2 parent studies was combined with the data from this study for the analysis of safety as planned.
Arm/Group | Bosutinib, CP1L | Bosutinib, CP2L | Bosutinib, CP3L/CP4L | Bosutinib, ADV | Bosutinib, Total
All-Cause Mortality (participants affected / at risk) | 23/248 | 55/284 | 30/119 | 98/167 | 206/818
Serious Adverse Events (participants affected / at risk) | 102/248 | 124/284 | 44/119 | 98/167 | 368/818
Other Adverse Events (participants affected / at risk) | 239/248 | 283/284 | 119/119 | 164/167 | 805/818
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib, CP1L (N=248) | Bosutinib, CP2L (N=284) | Bosutinib, CP3L/CP4L (N=119) | Bosutinib, ADV (N=167) | Bosutinib, Total (N=818)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 5 | 1 | 8 | 20
Anaemia (Blood and lymphatic system disorders) | 6 | 3 | 0 | 6 | 15
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 8 | 9
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 4 | 2 | 8
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 4
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 2
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Leukostasis syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 6 | 5 | 2 | 2 | 15
Cardiac failure congestive (Cardiac disorders) | 2 | 6 | 1 | 1 | 10
Atrial fibrillation (Cardiac disorders) | 1 | 4 | 3 | 1 | 9
Coronary artery disease (Cardiac disorders) | 3 | 2 | 2 | 1 | 8
Acute myocardial infarction (Cardiac disorders) | 1 | 3 | 1 | 2 | 7
Cardiac failure (Cardiac disorders) | 0 | 4 | 1 | 1 | 6
Pericarditis (Cardiac disorders) | 2 | 1 | 1 | 1 | 5
Angina pectoris (Cardiac disorders) | 0 | 3 | 1 | 0 | 4
Myocardial infarction (Cardiac disorders) | 0 | 0 | 3 | 1 | 4
Left ventricular dysfunction (Cardiac disorders) | 0 | 2 | 0 | 1 | 3
Angina unstable (Cardiac disorders) | 0 | 2 | 0 | 0 | 2
Pericardial haemorrhage (Cardiac disorders) | 0 | 2 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Cardiorenal syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 1 | 0 | 0 | 4
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Pleuropericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Cytogenetic abnormality (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 1 | 0 | 0 | 1
Glaucoma (Eye disorders) | 1 | 1 | 0 | 1 | 3
Cataract (Eye disorders) | 1 | 1 | 0 | 0 | 2
Visual impairment (Eye disorders) | 1 | 0 | 0 | 1 | 2
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 1
Retinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 1
Retinopathy hypertensive (Eye disorders) | 0 | 0 | 1 | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 8 | 1 | 4 | 22
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 0 | 5 | 11
Vomiting (Gastrointestinal disorders) | 3 | 2 | 0 | 5 | 10
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 6 | 8
Gastritis (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 6
Pancreatitis acute (Gastrointestinal disorders) | 1 | 3 | 0 | 1 | 5
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 4
Inguinal hernia (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 4
Pancreatitis (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 4
Colitis (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Gastric ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Mesenteric artery embolism (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Oesophageal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 8 | 8 | 2 | 11 | 29
Disease progression (General disorders) | 0 | 3 | 1 | 8 | 12
Chest pain (General disorders) | 1 | 3 | 0 | 4 | 8
General physical health deterioration (General disorders) | 0 | 1 | 0 | 6 | 7
Asthenia (General disorders) | 0 | 4 | 0 | 1 | 5
Pain (General disorders) | 1 | 0 | 0 | 2 | 3
Chills (General disorders) | 0 | 1 | 0 | 1 | 2
Death (General disorders) | 1 | 1 | 0 | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 2 | 2
Oedema (General disorders) | 0 | 0 | 1 | 1 | 2
Adhesion (General disorders) | 0 | 1 | 0 | 0 | 1
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 1
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 1
Swelling (General disorders) | 0 | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 4 | 0 | 1 | 7
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1 | 1 | 3
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 2 | 3
Gallbladder disorder (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Perforation bile duct (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 1 | 0 | 1 | 3
Anaphylactic shock (Immune system disorders) | 2 | 0 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 10 | 15 | 0 | 19 | 44
Sepsis (Infections and infestations) | 1 | 4 | 1 | 6 | 12
Cellulitis (Infections and infestations) | 3 | 3 | 1 | 1 | 8
Urinary tract infection (Infections and infestations) | 2 | 4 | 0 | 1 | 7
Bronchitis (Infections and infestations) | 2 | 3 | 1 | 0 | 6
Gastroenteritis (Infections and infestations) | 3 | 3 | 0 | 0 | 6
Influenza (Infections and infestations) | 0 | 4 | 1 | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 0 | 4
Appendicitis (Infections and infestations) | 1 | 1 | 1 | 0 | 3
Atypical pneumonia (Infections and infestations) | 1 | 2 | 0 | 0 | 3
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 3 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 2 | 1 | 0 | 3
Infection (Infections and infestations) | 1 | 2 | 0 | 0 | 3
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Device related infection (Infections and infestations) | 0 | 1 | 0 | 1 | 2
Erysipelas (Infections and infestations) | 0 | 2 | 0 | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0 | 0 | 2
Infectious pleural effusion (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Large intestine infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 2 | 0 | 0 | 2
Septic shock (Infections and infestations) | 0 | 1 | 0 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 2
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 1 | 2
Tooth abscess (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 1 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Catheter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Dengue fever (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Dermatitis infected (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Eczema infected (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Gingival abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Malaria (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Orchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pneumonia necrotising (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pulmonary mycosis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Salmonella bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Salmonellosis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 3
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 2
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Exposure during pregnancy (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Failure to anastomose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Traumatic lung injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Wound haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 8 | 1 | 0 | 0 | 9
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 0 | 0 | 5
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1 | 2
Lipase increased (Investigations) | 1 | 1 | 0 | 0 | 2
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 1
Intraocular pressure increased (Investigations) | 0 | 1 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 1
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 1 | 3 | 8
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 3
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 3
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 0 | 6
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Mandibular mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 2 | 6
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0 | 3
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1 | 3
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 2
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 2
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Bladder squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Follicle centre lymphoma, follicular grade I, II, III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 0 | 2 | 8 | 13
Syncope (Nervous system disorders) | 1 | 4 | 0 | 0 | 5
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 0 | 1 | 4
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2 | 0 | 2 | 4
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 2 | 3
Cerebral infarction (Nervous system disorders) | 0 | 2 | 0 | 1 | 3
Cerebellar infarction (Nervous system disorders) | 0 | 2 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 2
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 2
Seizure (Nervous system disorders) | 2 | 0 | 0 | 0 | 2
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Encephalitis post varicella (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Monoparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Dissociative disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 5 | 6 | 1 | 3 | 15
Renal failure (Renal and urinary disorders) | 1 | 2 | 1 | 1 | 5
Haematuria (Renal and urinary disorders) | 1 | 2 | 0 | 0 | 3
Calculus urinary (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 2
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
End stage renal disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 2
Breast hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 15 | 8 | 8 | 43
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 3 | 5 | 16
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2 | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 5 | 6
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0 | 4
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 3
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 8 | 1 | 1 | 11
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1 | 4
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Circumoral oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Pregnancy of partner (Social circumstances) | 2 | 0 | 1 | 0 | 3
Allogenic bone marrow transplantation therapy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 1
Cyst removal (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 2 | 0 | 1 | 4
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 2
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bosutinib, CP1L (N=248) | Bosutinib, CP2L (N=284) | Bosutinib, CP3L/CP4L (N=119) | Bosutinib, ADV (N=167) | Bosutinib, Total (N=818)
Thrombocytopenia (Blood and lymphatic system disorders) | 80 | 117 | 45 | 69 | 311
Anaemia (Blood and lymphatic system disorders) | 72 | 87 | 28 | 64 | 251
Neutropenia (Blood and lymphatic system disorders) | 35 | 46 | 23 | 35 | 139
Leukopenia (Blood and lymphatic system disorders) | 25 | 37 | 5 | 25 | 92
Diarrhoea (Gastrointestinal disorders) | 177 | 244 | 99 | 124 | 644
Nausea (Gastrointestinal disorders) | 89 | 132 | 58 | 78 | 357
Vomiting (Gastrointestinal disorders) | 88 | 106 | 47 | 72 | 313
Abdominal pain (Gastrointestinal disorders) | 39 | 77 | 28 | 34 | 178
Abdominal pain upper (Gastrointestinal disorders) | 40 | 59 | 21 | 16 | 136
Constipation (Gastrointestinal disorders) | 18 | 44 | 16 | 28 | 106
Dyspepsia (Gastrointestinal disorders) | 22 | 29 | 12 | 12 | 75
Toothache (Gastrointestinal disorders) | 14 | 19 | 5 | 3 | 41
Pyrexia (General disorders) | 50 | 79 | 17 | 59 | 205
Fatigue (General disorders) | 42 | 73 | 27 | 35 | 177
Asthenia (General disorders) | 26 | 45 | 10 | 19 | 100
Oedema peripheral (General disorders) | 17 | 32 | 13 | 18 | 80
Pain (General disorders) | 7 | 22 | 7 | 12 | 48
Oedema (General disorders) | 15 | 16 | 4 | 9 | 44
Chest pain (General disorders) | 7 | 21 | 4 | 11 | 43
Nasopharyngitis (Infections and infestations) | 30 | 40 | 14 | 9 | 93
Upper respiratory tract infection (Infections and infestations) | 39 | 32 | 12 | 10 | 93
Influenza (Infections and infestations) | 26 | 30 | 13 | 6 | 75
Urinary tract infection (Infections and infestations) | 15 | 31 | 7 | 2 | 55
Bronchitis (Infections and infestations) | 17 | 16 | 7 | 6 | 46
Alanine aminotransferase increased (Investigations) | 90 | 67 | 19 | 17 | 193
Aspartate aminotransferase increased (Investigations) | 74 | 59 | 10 | 17 | 160
Lipase increased (Investigations) | 52 | 29 | 8 | 9 | 98
Blood creatinine increased (Investigations) | 23 | 36 | 16 | 10 | 85
Weight decreased (Investigations) | 16 | 36 | 7 | 9 | 68
Amylase increased (Investigations) | 30 | 18 | 6 | 5 | 59
Blood creatine phosphokinase increased (Investigations) | 23 | 18 | 2 | 3 | 46
Blood alkaline phosphatase increased (Investigations) | 20 | 10 | 6 | 9 | 45
Decreased appetite (Metabolism and nutrition disorders) | 23 | 41 | 15 | 21 | 100
Hypophosphataemia (Metabolism and nutrition disorders) | 26 | 12 | 3 | 10 | 51
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 16 | 5 | 10 | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 32 | 55 | 21 | 24 | 132
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 43 | 15 | 16 | 100
Pain in extremity (Musculoskeletal and connective tissue disorders) | 23 | 35 | 10 | 19 | 87
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 26 | 6 | 14 | 62
Bone pain (Musculoskeletal and connective tissue disorders) | 11 | 20 | 9 | 11 | 51
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 11 | 12 | 9 | 44
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 14 | 8 | 7 | 43
Headache (Nervous system disorders) | 41 | 54 | 31 | 30 | 156
Dizziness (Nervous system disorders) | 25 | 26 | 18 | 21 | 90
Insomnia (Psychiatric disorders) | 12 | 10 | 10 | 15 | 47
Cough (Respiratory, thoracic and mediastinal disorders) | 32 | 70 | 26 | 33 | 161
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 25 | 34 | 13 | 30 | 102
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 26 | 32 | 20 | 14 | 92
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 37 | 11 | 13 | 76
Rash (Skin and subcutaneous tissue disorders) | 65 | 105 | 34 | 52 | 256
Pruritus (Skin and subcutaneous tissue disorders) | 20 | 29 | 20 | 10 | 79
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 22 | 8 | 4 | 44
Hypertension (Vascular disorders) | 24 | 30 | 10 | 11 | 75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT01903733/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/33/NCT01903733/SAP_001.pdf